CLINICAL TRIAL: NCT06665672
Title: Effect of Vibro-acoustic Stimulation on Night Shift Worker Sleep, Alertness, and Recovery (The Sleep Vibe Study)
Brief Title: Effect of a Wrist-worn Device That Produces a Small Vibration on Sleep and Performance That Can Occur During and After Night Shift Work
Acronym: Sleep-Vibe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Daniel Patterson, PhD, NRP (Other)
Responsible Party: Sponsor-Investigator, Daniel Patterson, PhD, NRP, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY24060106
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Sleep Duration; Psychomotor Performance
Keywords: Night shifts; Sleep duration; Nap; Shift work; Performance

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be blinded to the condition (arm) when the ApolloNeuro device is to be applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Apollo device applied followed by no device applied (Experimental): Participants will be randomized to first wear the Apollo Neuro device immediately before, during, and immediately after sleep opportunities during the study protocol. Next, the participant will complete the protocol without the device.
  Interventions: Device: Wrist worn vibro-acoustic device
- No device applied followed by the Apollo device applied (Experimental): Participants will be randomized to first complete the protocol without the Apollo Neuro device applied then complete a condition with the Apollo Neuro device applied immediately before, during, and immediately after sleep opportunities during the study protocol.
  Interventions: Device: Wrist worn vibro-acoustic device

INTERVENTIONS:
Device: Wrist worn vibro-acoustic device — The Apollo device is a wrist worn device that is similar to a typical wristwatch. It emits a vibration pattern based on settings selected on a designated mobile app.
  Other Names: Apollo

SUMMARY:
The overarching goal of this research study is to determine "proof of concept" of effect of a non-invasive sleep aid device on sleep and performance during sleep opportunities (naps) that occur during and after simulated night shift work.

Aim 1: To determine the effect of the ApolloNeuro device on sleep duration, sleep architecture, blood pressure, heart rate variability, and subjective ratings of sleep quality during and after simulated night shift work.

Aim 2: To determine the effect of the ApolloNeuro device on post-sleep psychomotor performance.

DETAILED DESCRIPTION:
Night shift workers suffer from poor sleep quality, high levels of fatigue, and irregular sleep patterns. The overarching goal of this research study is to determine "proof of concept" of effect of a non-invasive sleep aid device on sleep and performance during sleep opportunities (naps) that occur during and after simulated night shift work. The device is commercially available and worn on the wrist (the ApolloNeuro). We will use a laboratory-based, randomized crossover trial with two conditions tested. With 24 total subjects enrolled and 20 total completing the study as designed, we have 80% power to detect a moderate to large effect size difference between the two conditions tested. Study findings will guide a "go-no-go" decision for future, large-sample studies.

ELIGIBILITY:
Inclusion Criteria:

1. are 18 years of age or older;
2. have not been diagnosed or told by a healthcare clinician that they have a medical condition that may impact their blood pressure or cardiovascular health/system;
3. can abstain from smoking tobacco or chewing tobacco / nicotine products during the protocol and data collection;
4. can abstain from alcohol and moderate to high intensity exercise during the protocol and data collection;
5. are not prescribed medications or take over the counter medications that may impact blood pressure or heart rate (a team physician will review any reported medications identified during screening);
6. do not have a physical condition that may interfere with application of non-invasive devices on the wrist, upper arm, or chest for purposes of data collection with non-invasive devices;
7. feel that they can avoid working and complete the study protocol without interruption.
8. a public safety or healthcare shift worker based on standard licensing / certification requirements in the state of Pennsylvania.

Exclusion Criteria:

An individual will be excluded if they report:

1. a medical condition or diagnosis that may impact their blood pressure or heart rate;
2. taking any standing medications or prescriptions, other than over the counter medications or contraceptives, that may impact their blood pressure or heart rate;
3. are unable to adhere to the study protocol that involves abstaining from alcohol, tobacco products (nicotine), and moderate to intense exercise during the study protocol and data collection periods;
4. have a physical condition that may limit use of non-invasive devices applied to the wrist, upper arm, or chest for data collection purposes.
5. being pregnant.
6. "heavy" alcohol use as defined by the CDC (8 or more drinks per week in women or 15 or more drinks per week in men)?

Because participants will have their sleep interrupted during the in-lab sleep opportunity, it is important that staff and the study team know if the participant has ever experienced the following:

A] Sleep Paralysis; B] Night Terrors; C] Have Obstructive Sleep Apnea which requires the use of a CPAP Device; D] Become angry towards others when abruptly woken up; E] Become physical towards others when abruptly woken up.

Mild annoyance and feelings of fatigue or sleepiness with being woken by staff is expected and not a reason for exclusion in this research study.

Answering YES to any of the above (A-E) will result in a discussion with the study team physician to discuss with the individual and make a determination if the individual can or should participate in this research study.

All who voluntarily participate should be without significant health issues and without health concerns that may affect their blood pressure.

All who voluntarily participate should not be on medications that fall within the following categories:

A] Antihypertensives; B] Analgesics; C] Beta blockers; D] Diuretics; E] Stimulants; F] Sedatives; G] Steroids.

Participants must not take any medications with sedative effects or effects on sleep during the study protocol and data collection periods (such as NyQuil).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Mean sleep duration | Two time points examined. First, from the start of the simulated night shift 30-minute nap opportunity to the end at 30 minutes. Second, from the start of the recovery sleep period starting at 9am and ending at 2pm.
  Sleep duration is measured in minutes

SECONDARY OUTCOMES:
Mean number of lapses in psychomotor performance at 10 minutes after participants wake from sleep period | Measured at two time points. First, measured at 10 minutes after waking from the 30-minute nap opportunity during the simulated night shift. Second, measured at 10 minutes after participants wake from the 5-hour recovery sleep period..
  The 3-minute Psychomotor Vigilance Test Brief (PVT-B) is a reliable and valid measure of psychomotor performance. Investigators will assess the number of PVT-B Lapses for each participant measured at 10 minutes after waking from the 30-minute simulated shift nap opportunity. Number of Lapses is measured as a count and ranges from 0 to 50 or more during a single test.
Proportion with a dip in systolic blood pressure during 30-min nap opportunity that is greater than or equal to 10% | During the 30-min nap opportunity that occurs during the simulated 24-hour night shift
  The proportion of participants with a dip in systolic blood pressure (SBP) during the 30-min nap opportunity. SBP dipping - defined as - as ((mean wake hours SBP - mean sleep SBP divided by mean wake hours SBP) X 100). The percentage can range from 0 to 100.
Proportion with a dip in systolic blood pressure during the 5-hour recovery sleep period | During the 5-hour recovery sleep period that occurs after the 24-hour simulated night shift
  The proportion of participants with a dip in systolic blood pressure (SBP) during the 5-hour recovery sleep period. SBP dipping - defined as - ((mean wake hours SBP - mean sleep SBP divided by mean wake hours SBP) x 100). The percentage can range from 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Paul D Patterson, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified study data may be provided to researchers at the University of Pittsburgh, other institutions and/or federal repositories for the purposes of collaboration on the proposed research. Sharing will be completed under an approved sharing agreement.
Supporting Information: Study Protocol, ICF
Time Frame: December 2026
Access Criteria: Reviewed on a case by case basis